CLINICAL TRIAL: NCT03935308
Title: Phase I Study Of MR-guided Stereotactic Body Radiotherapy (SBRT) With Simultaneous Integrated Boost (SIB) To the Dominant Intraprostatic Lesion(s) (DILs) in Men With Localized Prostate Cancer
Brief Title: Phase I Study MR-guided SBRT to PCa
Acronym: MRgRTPCa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator left the institution.
Sponsor: Henry Ford Health System (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Stephen Brown, co-Lead, Translational Oncology Research, Henry Ford Cancer Institute, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRgSBRT
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Low or Intermediate Risk Prostate Cancer
Keywords: prostate cancer, MRI, intraprostatic lesions
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MR-guided SBRT With SIB to the DILs to Prostate Cancer (Experimental): Dose escalation to the DIL(s) will be performed in the traditional Phase I 3+3 design. Patients will be treated in four cohorts (three patients per dose level) starting with a dose of 9 Gy to the DIL(s). If no dose limiting toxicity (DLT), defined below, is observed after 90 days, then an additional three patients will be entered at the next dose level. Dose to the DIL(s) will be escalated at 1 Gy increments until DLT is observed or if maximum dose level (60 Gy in 5 fractions of 12 Gy) is reached with no observed DLT. If one of the three patients experience a DLT at a particular dose level an additional three patients will be enrolled at that level. If two or more patients experience a DLT a lower dose level will be explored to define the maximum tolerated dose (MTD). The three patients within any cohort can be enrolled simultaneously or sequentially without any waiting period among them.
  Interventions: Radiation: MR guided Linear Accelerator

INTERVENTIONS:
Radiation: MR guided Linear Accelerator — The aim is to perform treatment planning to compute the highest feasible simultaneous boosting dose to the intraprostatic lesion while respecting normal tissue dose constraints. Patients will be treated with MR-guided localization and adaptive planning techniques.

SUMMARY:
1) investigate the feasibility, tolerance, and safety of dose escalation via MR-guided stereotactic body radiation therapy and simultaneous integrated boost to the dominant intraprostatic lesions (DILs), 2) to assess the feasibility of DIL visualization based on multi-parametric MRI (mpMRI), and 3) to characterize longitudinal changes in imaging characteristics and identify urinary biomarkers for treatment response prediction

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma.
* Patients with low or favorable intermediate risk prostate cancer and patients with unfavorable intermediate risk prostate cancer who decline androgen deprivation therapy
* Pretreatment evaluations must be completed as specified in Section 4.0
* Patients must sign a study-specific informed consent form prior to study participation.
* No contraindication to MRI. For example, patients with metal fragments or implanted devices such as pacemakers and aneurysm clips may not be eligible for the study
* At least one intraprostatic lesion can be identified on the mpMR images.
* Patients agree to have hydrogel placed.

Exclusion Criteria:

* Patients who have a contraindication to contrast-enhanced MRI are not eligible. Patients with an implanted device such as a pacemaker or metal fragments are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose to DILs until dose limiting toxicity (>=3 grade 3 GI/GU toxicity) is observed or if maximum dose level is reached | 2 years
  The study aims to evaluate the safety and feasibility to employ a simultaneous integrated boost to MRI detected dominant intraprostatic lesion(s) during SBRT

SECONDARY OUTCOMES:
Quality of Life measures using the Epic questionnaire | 2 years
  Dose and volume data will be collected and correlated with treatment-related side effects and quality of life data.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dearnaley DP, Sydes MR, Graham JD, Aird EG, Bottomley D, Cowan RA, Huddart RA, Jose CC, Matthews JH, Millar J, Moore AR, Morgan RC, Russell JM, Scrase CD, Stephens RJ, Syndikus I, Parmar MK; RT01 collaborators. Escalated-dose versus standard-dose conformal radiotherapy in prostate cancer: first results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2007 Jun;8(6):475-87. doi: 10.1016/S1470-2045(07)70143-2. PMID 17482880
- [Background] Catton CN, Lukka H, Gu CS, Martin JM, Supiot S, Chung PWM, Bauman GS, Bahary JP, Ahmed S, Cheung P, Tai KH, Wu JS, Parliament MB, Tsakiridis T, Corbett TB, Tang C, Dayes IS, Warde P, Craig TK, Julian JA, Levine MN. Randomized Trial of a Hypofractionated Radiation Regimen for the Treatment of Localized Prostate Cancer. J Clin Oncol. 2017 Jun 10;35(17):1884-1890. doi: 10.1200/JCO.2016.71.7397. Epub 2017 Mar 15. PMID 28296582
- [Background] Pucar D, Hricak H, Shukla-Dave A, Kuroiwa K, Drobnjak M, Eastham J, Scardino PT, Zelefsky MJ. Clinically significant prostate cancer local recurrence after radiation therapy occurs at the site of primary tumor: magnetic resonance imaging and step-section pathology evidence. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):62-9. doi: 10.1016/j.ijrobp.2007.03.065. PMID 17707266
- [Background] Turkbey B, Mani H, Shah V, Rastinehad AR, Bernardo M, Pohida T, Pang Y, Daar D, Benjamin C, McKinney YL, Trivedi H, Chua C, Bratslavsky G, Shih JH, Linehan WM, Merino MJ, Choyke PL, Pinto PA. Multiparametric 3T prostate magnetic resonance imaging to detect cancer: histopathological correlation using prostatectomy specimens processed in customized magnetic resonance imaging based molds. J Urol. 2011 Nov;186(5):1818-24. doi: 10.1016/j.juro.2011.07.013. Epub 2011 Sep 25. PMID 21944089